CLINICAL TRIAL: NCT02999100
Title: A Randomized, Open-label Study to Characterize the Pharmacokinetics of Inhaled Oxytocin (GR121619) Compared With IM Oxytocin in Women in the Third Stage of Labour, and With IV Oxytocin in Non-pregnant, Non-lactating Women of Childbearing Potential
Brief Title: Comparison of Inhaled Oxytocin (IH) With Intramuscular (IM) Oxytocin in Pregnant Women and With Intravenous (IV) Oxytocin in Healthy Non-pregnant Women
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to reliably measure plasma oxytocin levels during third stage labour, regardless of administration method (intramuscular or inhaled).
Sponsor: GlaxoSmithKline (Industry)
Collaborators: InVentiv Clinique (Industry); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205920; 2016-002672-27 (EudraCT Number)
Record Dates: First submitted 2016-11-01; First posted 2016-12-21 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Postpartum Hemorrhage
Keywords: oxytocin; non-pregnant; pregnant; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 -IH oxytocin (Experimental): Women with an uncomplicated pregnancy in third stage of labour will be enrolled in the arm. Subjects will receive 400 micrograms (mcg) IH oxytocin. Subjects will be followed up in-person or via telephone within approximately 24 hr post dose and once between 7 days to 14 days
  Interventions: Drug: IH Oxytocin; Device: ROTAHALER
- Group 1 -IM oxytocin (Experimental): Women with an uncomplicated pregnancy in third stage of labour will be enrolled in the arm. Subjects will receive 10 I.U. IM oxytocin. Subjects will be followed up in-person or via telephone within approximately 24 hr post dose and once between 7 days to 14 days
  Interventions: Drug: IM Oxytocin
- Group 2 (IH and IV oxytocin) (Experimental): Group 2 will enrol healthy, non-pregnant, non-lactating female subjects of childbearing potential, and each subject will participate in 2 dosing sessions. Group 2 will be divided into two cohorts: Cohort A will enrol women on a combined oral contraceptive, and Cohort B will enrol women who are not using a hormonal form of contraceptive. Group 2 subjects will randomized to receive IH oxytocin, and IV oxytocin in a cross fashion. Subjects will be followed up in-person once between 7 days to 21 days
  Interventions: Drug: IH Oxytocin; Drug: IV Oxytocin; Device: ROTAHALER

INTERVENTIONS:
Drug: IH Oxytocin — Oxytocin will be supplied as colourless and clear hard capsule with powder blend for inhalation with unit dose strength 400 mcg and 200 mcg. It will be administered using ROTAHALER dry powder inhaler (DPI).
  Arms: Group 1 -IH oxytocin; Group 2 (IH and IV oxytocin)
Drug: IM Oxytocin — Oxytocin will be supplied for solution for infusion in 1ml ampoule containing colourless and clear sterile solution with unit dose strength 5 I.U./mL, or 10 I.U./mL for IM administration
  Arms: Group 1 -IM oxytocin
Drug: IV Oxytocin — Oxytocin will be supplied as solution for infusion in 1ml ampoule containing colourless and clear sterile solution to be administered as a 30-second IV bolus with unit dose strength 5 I.U./mL, or 10 I.U./mL.
  Arms: Group 2 (IH and IV oxytocin)
Device: ROTAHALER — ROTAHALER DPI device is a high airflow resistance capsule-based inhaler. It will be used to deliver IH oxytocin
  Arms: Group 1 -IH oxytocin; Group 2 (IH and IV oxytocin)

SUMMARY:
The study will evaluate a stable, dry-powder formulation of oxytocin, with the goal of reducing post-partum hemorrhage morbidity and mortality in resource poor settings. This study is being conducted to further assess safety and tolerability of inhaled oxytocin, and to characterize the drug levels of inhaled (IH) oxytocin when compared to oxytocin administered as standard of care. Two groups of subjects will be enrolled. Group 1 will enroll pregnant women, who will be randomized to receive either IH or intramuscular (IM) oxytocin as active management of the third stage of labour (after the baby is born). Group 2 will enroll non-pregnant women of childbearing potential, who will receive IH oxytocin and intravenous (IV) oxytocin in a cross over design over two dosing sessions This group will evaluate the safety and tolerability of IH and IV oxytocin.

ELIGIBILITY:
Inclusion Criteria:

All Groups:

* Between 18 and 40 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, and laboratory tests as required per protocol.
* Subject clinical chemistry and haematology values within an acceptable range for the population recruited and not of abnormal clinical significance. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor (if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Adequate peripheral venous access for cannulation.

Group 1 Only:

* Currently pregnant, with an uncomplicated pregnancy as determined by the investigator or designee.
* Estimated date of delivery within 24 weeks of screening.
* Planned spontaneous vaginal birth and considered by investigator at low risk for post partum hemorrhage (PPH).
* Planned birth in between the 37th and 42nd week of pregnancy.
* Women who qualify for oxytocin as appropriate for active management of TSL and who agree to have active management.

Group 2 Only:

* ECG normal, or abnormal and not clinically significant.
* FEV1 >80% of predicted.
* Systolic blood pressure >=90 millimeters of mercury (mmHg).
* Body mass index (BMI) within the range 18 - 32 Kilogram (kg)/square meter (m^2) (inclusive).
* Sex-Female.
* Group 2, Cohort A Only:

A female subject is eligible to participate if she is confirmed to be not pregnant at screening and on Day 1 (as confirmed by a negative serum or urine human chorionic gonadotrophin [hCG] test), not lactating, and the following condition applies:

Is of reproductive potential and agrees to use the same combined estrogen and progestogen oral contraceptive from 3 months prior to the first dose of study medication and until the follow-up contact.

This method of contraception is only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use their method of contraception

* Group 2, Cohort B Only:

A female subject is eligible to participate if she is confirmed to be not pregnant at screening and on Day 1 (as confirmed by a negative serum or urine hCG test), not lactating, and one of the following conditions applies:

Is of reproductive potential and has been using the same non-hormonal contraceptive method from 3 months prior to the first dose of study medication and until the follow-up contact.

Would be of reproductive potential, but has undergone bilateral tubal ligation or occlusion or bilateral salpingectomy at least 12 months prior to first dose of study medication.

Is of reproductive potential with only same sex partners or who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis, when this is their preferred and usual lifestyle. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

These methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use their method(s) of contraception.

Of Note: Group 2, Cohort B will enrol women of reproductive potential if they agree to use a nonhormonal contraceptive method from at least one month prior to receiving study drug and until the follow-up assessment. Although condoms with spermicide are not considered a highly effective method of contraception, the risk of receiving study drug during pregnancy is minimal for the following reasons:

Pregnancy testing must be negative at screening and on the first day of dosing. Dosing is completed no greater than 14 days from the start of dosing. Oxytocin has a well established rapid half-life. If a patient happened to conceive during the time of dosing, study drug would be eliminated before implantation would occur.

* All Groups: Capable of giving signed informed consent as described in Protocol which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

All Groups:

* Postmenopausal as defined by gynaecological history.
* Chronic lung condition of any etiology including asthma, Chronic obstructive pulmonary disease (COPD), emphysema, interstitial lung disease or active Tuberculosis (TB).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Blood pressure >140 systolic or >90 diastolic.

Group 1 Only:

* Females with planned Caesarean Section.
* Females with significant medical complications as determined by investigator.

Group 2 Only:

* Currently breastfeeding or lactating.
* QT duration corrected for heart rate by Fridericia's formula (QTcF) >450 milliseconds (msec).
* Alanine aminotransferase (ALT) and bilirubin >1.5 Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Subjects with highly-active or symptomatic gynaecological disorders (such as large symptomatic fibroids).

All Groups:

* Prescription or non-prescription drugs not approved by the investigator.
* Oxytocin for any reason (including, but not limited to, induction or augmentation of labour) prior to administration of study-related oxytocin.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 units. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 milliliter [ml]) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* Current smokers or subjects with a history of smoking within 6 months of screening, or with a total pack year history of >5 pack years. Confirmatory use via a Smokerlyzer is at the discretion of the local investigator, but is advised if the subject's recent smoking history is in doubt.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation (e.g. allergy to any previous inhaler use).
* Participation in another clinical trial, which in the opinion of the investigator, jeopardizes the subject's safety or study outcomes.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigation product within the following time period prior to the first dosing day in the current study: 30 days or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Group 2 Only:

* Presence of hepatitis B surface antigen or positive hepatitis C antibody test result.
* A positive Human Immunodeficiency Virus (HIV) antibody test.
* A positive pre-study drugs of abuse test (not explained by diet or approved concomitant medications).
* A positive alcohol breath test.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Clayton, Victoria, Australia
- United Kingdom (2):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Cambridge

REFERENCES:
- [Derived] Oliver VL, Siederer S, Cahn A, Gajewska-Knapik K, Gibson RA, Goodall C, Kirkpatrick C, Murray J, Nguyen TH, Schneider I, Lambert P, McIntosh MP, Parry S. Exploring the role of ex vivo metabolism on blood and plasma measurements of oxytocin among women in the third stage of labour: A post hoc study. Br J Clin Pharmacol. 2023 Dec;89(12):3669-3680. doi: 10.1111/bcp.15865. Epub 2023 Aug 24. PMID 37522415
- [Derived] Gajewska-Knapik K, Kumar S, Sutton-Cole A, Palmer KR, Cahn A, Gibson RA, Kirkpatrick C, Parry S, Schneider I, Siederer S, Stylianou A, Hacquoil K, Powell M, Ellis M, McIntosh MP, Lambert P. Pharmacokinetics and safety of inhaled oxytocin compared with intramuscular oxytocin in women in the third stage of labour: A randomized open-label study. Br J Clin Pharmacol. 2023 Dec;89(12):3681-3689. doi: 10.1111/bcp.15860. Epub 2023 Aug 31. PMID 37485589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 2 part study: Part 1 enrolled pregnant women, randomized to receive either inhaled (IH) or intramuscular (IM) oxytocin as active management of the third stage of labor. Part 2 enrolled non-pregnant women of childbearing potential and received IH oxytocin and intravenous (IV) oxytocin in a cross over design.
Pre-assignment Details: A total of 31 participants were enrolled in the study. This study was terminated due to inability to reliably measure plasma oxytocin levels in women in third stage labor, regardless of administration method (IH, IM or IV).
Groups:
- 400 mcg Oxytocin IH: Participants with uncomplicated pregnancy received 400 micrograms (mcg) IH oxytocin during third stage of labor (within 5 minutes of birth) via ROTAHALER dry powder inhaler (DPI). Participants were followed up in-person or via telephone within approximately 24 hours post dose and once between 7 days to 14 days.
- 17 mcg Oxytocin IM: Participants with uncomplicated pregnancy received 17 mcg IM oxytocin injection during third stage of labor (within 5 minutes of birth) in the anterior shoulder. Participants were followed up in-person or via telephone within approximately 24 hours post dose and once between 7 days to 14 days.
- Contraceptives+400 mcg Oxytocin IH, Then 8.5mcg Oxytocin IV: Healthy participants of childbearing potential were administered oral contraceptive along with 400 mcg oxytocin IH during Session 1 and received 8.5 mcg oxytocin IV during Session 2. Participants were followed up in-person or via telephone within 7 days and no greater than 21 days after last study drug administration.
- Contraceptives+8.5mcg Oxytocin IV, Then 400 mcg Oxytocin IH: Healthy participants of childbearing potential were administered oral contraceptives along with 8.5 mcg oxytocin IV during Session 1 and received 400 mcg oxytocin IH during Session 2. Participants were followed up in-person or via telephone within 7 days and no greater than 21 days after last study drug administration.
- 400 mcg Oxytocin IH, Then 8.5 mcg Oxytocin IV: Healthy participants of childbearing potential were administered 400 mcg oxytocin IH during Session 1 and received 8.5 mcg oxytocin IV during Session 2. Participants were followed up in-person or via telephone within 7 days and no greater than 21 days after last study drug administration.
- 8.5 mcg Oxytocin IV, Then 400 mcg Oxytocin IH: Healthy participants of childbearing potential were administered 8.5 mcg oxytocin IV during Session 1 and received 400 mcg oxytocin IH during Session 2. Participants were followed up in-person or via telephone within 7 days and no greater than 21 days after last study drug administration.
Period: Part 1 (up to 15 Days)
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM | Contraceptives+400 mcg Oxytocin IH, Then 8.5mcg Oxytocin IV | Contraceptives+8.5mcg Oxytocin IV, Then 400 mcg Oxytocin IH | 400 mcg Oxytocin IH, Then 8.5 mcg Oxytocin IV | 8.5 mcg Oxytocin IV, Then 400 mcg Oxytocin IH
Started | 9 | 8 | 0 | 0 | 0 | 0
Completed | 9 | 7 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2 (Day 1): Dosing Session 1
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM | Contraceptives+400 mcg Oxytocin IH, Then 8.5mcg Oxytocin IV | Contraceptives+8.5mcg Oxytocin IV, Then 400 mcg Oxytocin IH | 400 mcg Oxytocin IH, Then 8.5 mcg Oxytocin IV | 8.5 mcg Oxytocin IV, Then 400 mcg Oxytocin IH
Started | 0 (Participants from Part 1 did not enter Part 2) | 0 (Participants from Part 1 did not enter Part 2) | 5 (New participants were enrolled in Part 2 of study) | 3 (New participants were enrolled in Part 2 of study) | 3 (New participants were enrolled in Part 2 of study) | 3 (New participants were enrolled in Part 2 of study)
Completed | 0 | 0 | 4 | 3 | 3 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2 (Day 14): Dosing Session 2
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM | Contraceptives+400 mcg Oxytocin IH, Then 8.5mcg Oxytocin IV | Contraceptives+8.5mcg Oxytocin IV, Then 400 mcg Oxytocin IH | 400 mcg Oxytocin IH, Then 8.5 mcg Oxytocin IV | 8.5 mcg Oxytocin IV, Then 400 mcg Oxytocin IH
Started | 0 | 0 | 4 | 3 | 3 | 2
Completed | 0 | 0 | 4 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM | Contraceptives+400 mcg Oxytocin IH, Then 8.5mcg Oxytocin IV | Contraceptives+8.5mcg Oxytocin IV, Then 400 mcg Oxytocin IH | 400 mcg Oxytocin IH, Then 8.5 mcg Oxytocin IV | 8.5 mcg Oxytocin IV, Then 400 mcg Oxytocin IH | Total
Number analyzed (Participants) | 9 | 8 | 5 | 3 | 3 | 3 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (3.49) | 28.1 (5.84) | 24.0 (4.53) | 30.7 (0.58) | 37.3 (1.53) | 27.7 (6.66) | 29.6 (5.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 5 | 3 | 3 | 3 | 31
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian - South East Asian Heritage | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White - White/Caucasian/European Heritage | 7 | 5 | 4 | 3 | 3 | 3 | 25
  Asian - Central/South Asian Heritage | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Mixed race | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Plasma Concentration Time Profile of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate concentration of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Predose, 3 minutes, 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 2.5 hours, 3 hours and 4 hours post dose Day 1
Population: Pharmacokinetic Population includes all participants in Safety population for whom a pharmacokinetic sample was obtained & analysed.Safety Population includes participants who received at least one dose of study medication.Only those participants with data available at specified data points were analyzed (represented by n= X in the category titles)
Measure: Median (Full Range); unit: Picograms per milliliter
Groups:
- 400 mcg Oxytocin IH: Participants with uncomplicated pregnancy received 400 micrograms (mcg) IH oxytocin during third stage of labo (within 5 minutes of birth) via ROTAHALER dry powder inhaler (DPI). Participants were followed up in-person or via telephone within approximately 24 hours post dose and once between 7 days to 14 days.
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Picograms per milliliter
  Pre-dose; n=9, 8 | 0.000 [0.00 to 5.32] | 0.000 [0.00 to 0.00]
  3 minutes post dose; n= 7, 7: number analyzed (Participants) | 7 | 7
  3 minutes post dose; n= 7, 7 | 0.000 [0.00 to 33.54] | 0.000 [0.00 to 0.00]
  5 minutes post dose; n=8, 7: number analyzed (Participants) | 8 | 7
  5 minutes post dose; n=8, 7 | 1.020 [0.00 to 35.96] | 0.000 [0.00 to 4.35]
  10 minutes post dose; n=7, 8: number analyzed (Participants) | 7 | 8
  10 minutes post dose; n=7, 8 | 0.000 [0.00 to 24.58] | 0.000 [0.00 to 4.50]
  15 minutes post dose; n=8, 8: number analyzed (Participants) | 8 | 8
  15 minutes post dose; n=8, 8 | 0.000 [0.00 to 13.67] | 0.000 [0.00 to 3.61]
  20 minutes post dose; n=8, 6: number analyzed (Participants) | 8 | 6
  20 minutes post dose; n=8, 6 | 0.000 [0.00 to 8.70] | 0.000 [0.00 to 3.19]
  30 minutes post dose; n=8, 7: number analyzed (Participants) | 8 | 7
  30 minutes post dose; n=8, 7 | 0.000 [0.00 to 8.46] | 0.000 [0.00 to 3.53]
  1 hour post dose; n=8, 7: number analyzed (Participants) | 8 | 7
  1 hour post dose; n=8, 7 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 2.84]
  2 hours post dose; n=9, 7: number analyzed (Participants) | 9 | 7
  2 hours post dose; n=9, 7 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  2.5 hours post dose; n=9, 7: number analyzed (Participants) | 9 | 7
  2.5 hours post dose; n=9, 7 | 0.000 [0.00 to 3.54] | 0.000 [0.00 to 0.00]
  3 hours post dose; n=8, 7: number analyzed (Participants) | 8 | 7
  3 hours post dose; n=8, 7 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  4 hours post dose; n=8, 7: number analyzed (Participants) | 8 | 7
  4 hours post dose; n=8, 7 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

2. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate Cmax of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Picograms per milliliter
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Picograms per milliliter | 2.460 [NA to 35.96] — NA indicates that lower range could not be calculated due to high proportion of non-quantifiable [NQ] values (more than 50% of values were imputed i.e., NQ assigned zero concentration) which affected the calculation. | NA [NA to 4.50] — NA indicates that median and lower range could not be calculated due to high proportion of non-quantifiable [NQ] values (more than 50% of values were imputed i.e., NQ assigned zero concentration) which affected the calculation.

3. Primary Outcome: Part 1: Observed Plasma Concentration (Cp) 10 of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate observed plasma concentration of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: 10 minutes post dose Day 1
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Picogram per milliliter | NA [NA to 24.58] — NA indicates that median and lower range could not be calculated as values at specified time points (10 minutes post-dose) were below the limit of quantification. | NA [NA to 4.50] — NA indicates that median and lower range could not be calculated as values at specified time points (10 minutes post-dose) were below the limit of quantification.

4. Primary Outcome: Part 1: Observed Plasma Concentration (Cp) 20 of Oxytocin
Description: as for outcome 3
Time Frame: 20 minutes post dose Day 1
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Picogram per milliliter | NA [NA to 8.70] — NA indicates that median and lower range could not be calculated as values at specified time points (20 minutes post-dose) were below the limit of quantification. | 1.960 [NA to 3.19] — NA indicates that lower range could not be calculated as values at specified time points (20 minutes post-dose) were below the limit of quantification.

5. Primary Outcome: Part 1: Observed Plasma Concentration (Cp) 30 of Oxytocin
Description: as for outcome 3
Time Frame: 30 minutes post dose Day 1
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Picogram per milliliter | NA [NA to 8.46] — NA indicates that median and lower range could not be calculated as values at specified time points (30 minutes post-dose) were below the limit of quantification. | NA [NA to 3.53] — NA indicates that median and lower range could not be calculated as values at specified time points (30 minutes post-dose) were below the limit of quantification.

6. Primary Outcome: Part 1: Time to Reach Maximum Observed Concentration (Tmax) of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate Tmax of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 6 | 3
Hours | 0.15000 [0.0500 to 2.5000] | 0.25000 [0.1667 to 0.4833]

7. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate AUC (0-t) of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Predose, 3 minutes, 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 2.5 hours, 3 hours and 4 hours post dose on Day 1
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hour*picogram per milliliter
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Hour*picogram per milliliter | NA [NA to 8.1] — NA indicates that median and lower range could not be calculated due to high proportion of non-quantifiable [NQ] values (more than 50% of values were imputed i.e., NQ assigned zero concentration) which affected the calculation. | NA [NA to 2.3] — NA indicates that median and lower range could not be calculated due to high proportion of non-quantifiable [NQ] values (more than 50% of values were imputed i.e., NQ assigned zero concentration) which affected the calculation.

8. Primary Outcome: Part 1: Terminal Phase Half-life (t1/2) of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate t1/2 of oxytocin.
Time Frame: as for outcome 7
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Hours | NA [NA to NA] — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification. | NA [NA to NA] — NA indicates that data could not be calculated as all values in terminal elimination phase were below the limit of quantification.

9. Primary Outcome: Part 2: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. As SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. Safety Population includes participants who received at least one dose of study medication.
Time Frame: Up to 37 days
Population: Safety Population. Participants analysed (25) is greater than the number participants (14) started in Part 2 because Part 2 is a crossover design and participants were considered for 2 dosing sessions.
Measure: Count of Participants; unit: Participants
Groups:
- Combined Oral Contraceptives+400 mcg Oxytocin IH: Healthy participants of childbearing potential receiving oral contraceptive along with 400 mcg oxytocin IH.
- Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus: Healthy participants of childbearing potential receiving oral contraceptive along with 8.5 mcg oxytocin IV bolus. When the duration of IV oxytocin administered was less than or equal to 2 minutes then the IV dose administered was classified as an IV Bolus.
- Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion: Healthy participants of childbearing potential receiving oral contraceptive along with 8.5 mcg oxytocin IV.
- Non-Combined Oral Contraceptives+400 mcg Oxytocin IH: Healthy participants of childbearing potential using a non-hormonal form of contraception along with 400 mcg oxytocin IH.
- Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus: Healthy participants of childbearing potential using a non-hormonal form of contraception along with 8.5 mcg oxytocin IV bolus. When the duration of IV oxytocin administered was less than or equal to 2 minutes then the IV dose administered was classified as an IV Bolus.
- Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion: Healthy participants of childbearing potential using a non-hormonal form of contraception along with 8.5 mcg oxytocin IV.
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Participants
  Any non-SAE | 7 | 5 | 1 | 3 | 1 | 5
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part 2: Absolute Values of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour and 4 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Millimeters of mercury
  SBP: Pre-dose | 107.1 (5.24) | 116.0 (12.73) | 102.0 (5.66) | 105.4 (10.11) | 99.0 (NA) — NA indicates that standard deviation (SD) could not be calculated for a single participant | 107.2 (6.61)
  SBP: 5 minutes | 114.0 (6.16) | 118.2 (9.76) | 103.5 (9.19) | 108.4 (10.71) | 104.0 (NA) — NA indicates that SD could not be calculated for a single participant | 110.6 (15.14)
  SBP: 15 minutes | 108.9 (3.29) | 114.6 (9.40) | 106.0 (5.66) | 106.4 (9.50) | 98.0 (NA) — NA indicates that SD could not be calculated for a single participant | 106.0 (10.07)
  SBP: 30 minutes | 109.6 (4.04) | 111.2 (6.87) | 107.0 (8.49) | 113.2 (12.05) | 100.0 (NA) — NA indicates that SD could not be calculated for a single participant | 104.6 (10.95)
  SBP: 1 hour | 104.9 (6.26) | 111.4 (5.37) | 103.5 (2.12) | 108.8 (8.64) | 98.0 (NA) — NA indicates that SD could not be calculated for a single participant | 109.0 (12.61)
  SBP: 4 hours | 106.9 (5.11) | 111.4 (11.28) | 106.5 (3.54) | 102.0 (9.41) | 93.0 (NA) — NA indicates that SD could not be calculated for a single participant | 106.4 (3.21)
  DBP: Pre-dose | 65.1 (5.93) | 62.4 (7.54) | 67.0 (1.41) | 62.0 (6.36) | 58.0 (NA) — NA indicates that SD could not be calculated for a single participant | 64.2 (8.29)
  DBP: 5 minutes | 67.1 (7.67) | 67.0 (8.15) | 61.5 (7.78) | 65.2 (3.03) | 67.0 (NA) — NA indicates that SD could not be calculated for a single participant | 60.4 (5.68)
  DBP: 15 minutes | 65.4 (5.62) | 64.8 (7.43) | 65.5 (4.95) | 65.6 (3.36) | 68.0 (NA) — NA indicates that SD could not be calculated for a single participant | 62.4 (5.77)
  DBP: 30 minutes | 68.3 (6.07) | 65.2 (3.11) | 66.5 (4.95) | 69.6 (6.73) | 70.0 (NA) — NA indicates that SD could not be calculated for a single participant | 63.0 (5.48)
  DBP: 1 hour | 65.9 (4.85) | 65.8 (3.56) | 69.0 (5.66) | 66.6 (2.41) | 65.0 (NA) — NA indicates that SD could not be calculated for a single participant | 66.4 (9.21)
  DBP: 4 hours | 66.4 (7.57) | 61.6 (6.99) | 64.5 (9.19) | 60.0 (6.52) | 62.0 (NA) — NA indicates that SD could not be calculated for a single participant | 59.2 (5.07)

11. Primary Outcome: Part 2: Change From Baseline in SBP and DBP
Description: SBP and DBP of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Baseline was defined as the latest pre-dose assessment with a non-missing value at Day 1 (Pre-dose). Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), 5 minutes, 15 minutes, 30 minutes, 1 hour and 4 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Millimeters of mercury
  SBP: 5 minutes | 6.9 (6.47) | 2.2 (13.42) | 1.5 (3.54) | 3.0 (10.42) | 5.0 (NA) — NA indicates that SD could not be calculated for a single participant | 3.4 (10.88)
  SBP: 15 minutes | 1.7 (3.25) | -1.4 (14.67) | 4.0 (0.00) | 1.0 (11.02) | -1.0 (NA) — NA indicates that SD could not be calculated for a single participant | -1.2 (6.98)
  SBP: 30 minutes | 2.4 (2.07) | -4.8 (13.35) | 5.0 (2.83) | 7.8 (12.56) | 1.0 (NA) — NA indicates that SD could not be calculated for a single participant | -2.6 (7.80)
  SBP: 1 hour | -2.3 (4.27) | -4.6 (14.10) | 1.5 (3.54) | 3.4 (13.54) | -1.0 (NA) — NA indicates that SD could not be calculated for a single participant | 1.8 (9.71)
  SBP: 4 hours | -0.3 (3.82) | -4.6 (13.79) | 4.5 (2.12) | -3.4 (9.29) | -6.0 (NA) — NA indicates that SD could not be calculated for a single participant | -0.8 (7.95)
  DBP: 5 minutes | 2.0 (10.69) | 4.6 (3.58) | -5.5 (9.19) | 3.2 (6.46) | 9.0 (NA) — NA indicates that SD could not be calculated for a single participant | -3.8 (3.35)
  DBP: 15 minutes | 0.3 (6.92) | 2.4 (7.70) | -1.5 (6.36) | 3.6 (4.28) | 10.0 (NA) — NA indicates that SD could not be calculated for a single participant | -1.8 (5.50)
  DBP: 30 minutes | 3.1 (7.88) | 2.8 (8.04) | -0.5 (6.36) | 7.6 (9.94) | 12.0 (NA) — NA indicates that SD could not be calculated for a single participant | -1.2 (4.87)
  DBP: 1 hour | 0.7 (3.35) | 3.4 (6.54) | 2.0 (7.07) | 4.6 (3.97) | 7.0 (NA) — NA indicates that SD could not be calculated for a single participant | 2.2 (2.95)
  DBP: 4 hours | 1.3 (8.20) | -0.8 (4.97) | -2.5 (10.61) | -2.0 (3.24) | 4.0 (NA) — NA indicates that SD could not be calculated for a single participant | -5.0 (6.63)

12. Primary Outcome: Part 2: Change From Baseline in Heart Rate
Description: Heart rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Baseline was defined as the latest pre-dose assessment with a non-missing value at Day 1 (Pre-dose). Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), 5 minutes, 15 minutes, 30 minutes, 1 hour and 4 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Beats per minute
  5 minutes | 2.9 (6.99) | 13.8 (11.86) | 19.5 (3.54) | 7.4 (13.05) | -7.0 (NA) — NA indicates that SD could not be calculated for a single participant | 13.0 (7.52)
  15 minutes | 2.9 (11.51) | 4.4 (9.4) | 7 (7.07) | 2.6 (12.44) | -7.0 (NA) — NA indicates that SD could not be calculated for a single participant | 0.6 (3.29)
  30 minutes | -1.9 (7.29) | 1.2 (11.34) | 1 (1.41) | -3.6 (11.74) | -9.0 (NA) — NA indicates that SD could not be calculated for a single participant | -0.2 (4.09)
  1 hour | -5.9 (7.15) | 2.2 (8.56) | 4.5 (6.36) | -1.4 (10.04) | -10.0 (NA) — NA indicates that SD could not be calculated for a single participant | 0.2 (3.96)
  4 hours | 3.1 (6.49) | 5.8 (11.5) | 9 (22.63) | 6.2 (5.4) | -6.0 (NA) — NA indicates that SD could not be calculated for a single participant | 5.8 (3.49)

13. Primary Outcome: Part 2: Absolute Values of Heart Rate
Description: Heart rate was measured in semi-supine position after 5 minutes rest
Time Frame: Pre dose, 5 minutes, 15 minutes, 30 minutes, 1 hour and 4 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Beats per minute
  Pre dose | 71.1 (15.29) | 65.2 (5.93) | 63.5 (21.92) | 65 (9.3) | 81.0 (NA) — NA indicates that SD could not be calculated for a single participant | 63.6 (13.46)
  5 minutes | 74.0 (15.01) | 79 (8.15) | 83 (18.38) | 72.4 (14.1) | 74.0 (NA) — NA indicates that SD could not be calculated for a single participant | 76.6 (18.5)
  15 minutes | 74.0 (10.31) | 69.6 (5.64) | 70.5 (14.85) | 67.6 (11.93) | 74.0 (NA) — NA indicates that SD could not be calculated for a single participant | 64.2 (16.3)
  30 minutes | 69.3 (9.32) | 66.4 (6.47) | 64.5 (23.33) | 61.4 (7.96) | 72.0 (NA) — NA indicates that SD could not be calculated for a single participant | 63.4 (13.22)
  1 hour | 65.3 (10.59) | 67.4 (4.67) | 68 (15.56) | 63.6 (11.24) | 71.0 (NA) — NA indicates that SD could not be calculated for a single participant | 63.8 (13.12)
  4 hours | 74.3 (13.21) | 71 (5.7) | 72.5 (0.71) | 71.2 (5.54) | 75.0 (NA) — NA indicates that SD could not be calculated for a single participant | 69.4 (15.11)

14. Primary Outcome: Part 2: Absolute Values of PR Interval, QRS Duration, Corrected QT Interval Using Bazett's (QTcB) Formula and Corrected QT Interval Using Fredericia's Formula (QTcF) Interval
Description: Triplicate 12-lead electrocardiograms (ECGs) were recorded pre-dose and post-dose with participant in semi-supine position after 5 minutes rest. At each time point ECG was taken using an ECG machine that automatically measured PR interval, QRS duration, QTcB interval, and QTcF interval.
Time Frame: Pre-dose, 2 minutes, 10 minutes, 20 minutes, 30 minutes, 1 hour and 4 hours post dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Milliseconds
  PR interval: Pre-dose | 150.9 (23.67) | 156.0 (22.17) | 146.5 (21.92) | 139.8 (23.67) | 127.0 (NA) — NA indicates that SD could not be calculated for a single participant | 139.6 (28.32)
  PR interval: 2 minutes | 144.6 (25.36) | 158.4 (24.13) | 146.5 (14.85) | 140.0 (27.70) | 125.0 (NA) — NA indicates that SD could not be calculated for a single participant | 147.0 (30.36)
  PR interval: 10 minutes | 150.9 (27.90) | 161.6 (24.77) | 143.0 (21.21) | 146.2 (28.65) | 128.0 (NA) — NA indicates that SD could not be calculated for a single participant | 146.0 (31.96)
  PR interval: 20 minutes | 152.1 (29.59) | 161.2 (26.40) | 143.5 (20.51) | 147.4 (28.61) | 125.0 (NA) — NA indicates that SD could not be calculated for a single participant | 151.0 (32.08)
  PR interval: 30 minutes | 151.4 (28.96) | 158.8 (25.03) | 147.0 (14.14) | 146.0 (24.37) | 128.0 (NA) — NA indicates that SD could not be calculated for a single participant | 151.8 (30.43)
  PR interval: 1 hour | 154.4 (28.92) | 160.4 (22.88) | 147.5 (13.44) | 146.8 (27.65) | 129.0 (NA) — NA indicates that SD could not be calculated for a single participant | 150.0 (28.24)
  PR interval: 4 hours | 153.1 (23.43) | 155.8 (25.80) | 145.5 (16.26) | 141.6 (21.09) | 117.0 (NA) — NA indicates that SD could not be calculated for a single participant | 139.4 (29.37)
  QRS duration: Pre-dose | 91.4 (8.20) | 89.0 (5.52) | 99.0 (7.07) | 91.4 (8.85) | 94.0 (NA) — NA indicates that SD could not be calculated for a single participant | 89.0 (9.85)
  QRS duration: 2 minutes | 92.7 (7.11) | 89.4 (5.68) | 104.0 (4.24) | 90.4 (9.32) | 91.0 (NA) — NA indicates that SD could not be calculated for a single participant | 86.8 (6.26)
  QRS duration: 10 minutes | 92.3 (11.01) | 91.2 (5.67) | 98.5 (9.19) | 91.2 (9.18) | 91.0 (NA) — NA indicates that SD could not be calculated for a single participant | 89.2 (9.58)
  QRS duration: 20 minutes | 90.7 (8.96) | 87.8 (4.15) | 91.0 (18.38) | 90.2 (9.55) | 92.0 (NA) — NA indicates that SD could not be calculated for a single participant | 89.0 (11.92)
  QRS duration: 30 minutes | 91.3 (9.27) | 89.2 (5.22) | 100.0 (0.00) | 93.4 (8.88) | 93.0 (NA) — NA indicates that SD could not be calculated for a single participant | 92.2 (10.62)
  QRS: 1 hour | 90.9 (8.15) | 89.6 (4.83) | 99.0 (1.41) | 93.2 (9.34) | 91.0 (NA) — NA indicates that SD could not be calculated for a single participant | 89.4 (8.88)
  QRS: 4 hours | 92.3 (9.52) | 88.6 (3.21) | 106.0 (8.49) | 89.0 (6.04) | 92.0 (NA) — NA indicates that SD could not be calculated for a single participant | 90.0 (6.60)
  QTcF: Pre-dose | 401.7 (11.84) | 406.0 (19.51) | 406.5 (7.78) | 413.8 (12.15) | 416.0 (NA) — NA indicates that SD could not be calculated for a single participant | 411.6 (9.63)
  QTcF: 2 minutes | 403.0 (22.02) | 422.6 (21.51) | 432.5 (20.51) | 420.6 (12.50) | 426.0 (NA) — NA indicates that SD could not be calculated for a single participant | 427.4 (19.30)
  QTcF: 10 minutes | 407.0 (11.18) | 430.2 (20.23) | 413.5 (13.44) | 422.6 (13.15) | 421.0 (NA) — NA indicates that SD could not be calculated for a single participant | 412.8 (8.96)
  QTcF: 20 minutes | 407.0 (14.87) | 415.2 (26.22) | 419.5 (16.26) | 422.0 (8.28) | 408.0 (NA) — NA indicates that SD could not be calculated for a single participant | 416.6 (16.29)
  QTcF: 30 minutes | 406.4 (13.96) | 420.2 (15.96) | 411.0 (19.80) | 424.6 (8.20) | 413.0 (NA) — NA indicates that SD could not be calculated for a single participant | 417.0 (15.25)
  QTcF: 1 hour | 408.3 (11.90) | 416.0 (20.76) | 422.5 (0.71) | 420.2 (5.22) | 418.0 (NA) — NA indicates that SD could not be calculated for a single participant | 416.2 (18.57)
  QTcF: 4 hours | 410.4 (10.63) | 409.2 (17.63) | 420.5 (2.12) | 408.2 (22.92) | 410.0 (NA) — NA indicates that SD could not be calculated for a single participant | 415.6 (12.54)
  QTcB: Pre-dose | 413.2 (20.41) | 408.8 (24.01) | 413.8 (26.37) | 420.4 (16.10) | 441.7 (NA) — NA indicates that SD could not be calculated for a single participant | 418.4 (17.24)
  QTcB: 2 minutes | 422.3 (30.97) | 453.4 (26.42) | 464.4 (8.95) | 443.1 (20.62) | 460.9 (NA) — NA indicates that SD could not be calculated for a single participant | 453.5 (30.42)
  QTcB: 10 minutes | 421.3 (16.19) | 443.8 (22.71) | 429.0 (1.98) | 434.1 (25.91) | 439.1 (NA) — NA indicates that SD could not be calculated for a single participant | 421.7 (18.96)
  QTcB: 20 minutes | 416.0 (20.89) | 421.8 (29.04) | 425.5 (2.54) | 432.9 (17.19) | 418.4 (NA) — NA indicates that SD could not be calculated for a single participant | 418.9 (21.93)
  QTcB: 30 minutes | 415.1 (22.11) | 427.8 (19.67) | 415.1 (7.05) | 431.6 (18.64) | 423.9 (NA) — NA indicates that SD could not be calculated for a single participant | 419.6 (27.77)
  QTcB: 1 hour | 415.9 (15.66) | 419.5 (24.53) | 435.4 (13.98) | 423.2 (15.57) | 436.7 (NA) — NA indicates that SD could not be calculated for a single participant | 419.9 (25.24)
  QTcB: 4 hours | 422.4 (13.29) | 415.5 (15.04) | 439.0 (7.14) | 421.9 (28.51) | 429.3 (NA) — NA indicates that SD could not be calculated for a single participant | 426.4 (17.82)

15. Primary Outcome: Part 2: Number of Participants With Abnormal Respiratory Events
Description: Number of participants with abnormal respiratory events has been presented
Time Frame: Up to Day 37
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Participants | 2 | 1 | 0 | 0 | 0 | 0

16. Primary Outcome: Part 2: Forced Expiratory Volume at 1 Minute (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 measurements were taken electronically by spirometry on Day 1. At each time point, three best measurements were recorded.
Time Frame: Pre dose and 1 hour post dose on Day1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Liters
  Pre-dose | 3.251 (0.3125) | 3.440 (0.3121) | 3.130 (0.0707) | 3.384 (0.3051) | 3.630 (NA) — NA indicates that SD could not be calculated for a single participant | 3.284 (0.3488)
  1 hour | 3.184 (0.2769) | 3.374 (0.2964) | 3.110 (0.1980) | 3.306 (0.2874) | 3.380 (NA) — NA indicates that SD could not be calculated for a single participant | 3.190 (0.3768)

17. Primary Outcome: Part 2: Percent Oxygen in Blood
Description: Percent oxygen in blood was measured using pulse oximetry in a semi-supine position after 5 minutes rest. Pulse oximeter is a device that measures oxygen saturation of arterial blood in participants by utilizing a sensor attached typically to a finger, toe, or ear to determine the percentage of oxyhemoglobin in blood pulsating through a network of capillaries
Time Frame: Pre dose, 5 minutes, 15 minutes, 30 minutes, 1 hour and 4 hours post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of oxygen
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Percentage of oxygen
  Pre dose | 98.6 (1.4) | 99.4 (0.89) | 99.0 (1.41) | 97.2 (0.84) | 98.0 (NA) — NA indicates that SD could not be calculated for a single participant | 97.4 (0.89)
  5 minutes | 98.9 (1.21) | 99.0 (1.00) | 99.0 (1.41) | 98.0 (1.41) | 98.0 (NA) — NA indicates that SD could not be calculated for a single participant | 98.8 (1.30)
  15 minutes | 98.7 (1.25) | 98.8 (0.84) | 99.5 (0.71) | 97.8 (1.10) | 98.0 (NA) — NA indicates that SD could not be calculated for a single participant | 98.4 (1.14)
  30 minutes | 98.9 (0.9) | 98.4 (1.14) | 99.5 (0.71) | 98.2 (0.84) | 98.0 (NA) — NA indicates that SD could not be calculated for a single participant | 98.2 (1.10)
  1 hour | 98.4 (1.27) | 98.2 (1.3) | 99.0 (1.41) | 98 (0.71) | 99.0 (NA) — NA indicates that SD could not be calculated for a single participant | 98.2 (1.10)
  4 hours | 99.0 (0.82) | 98.4 (0.89) | 99.5 (0.71) | 97.8 (0.84) | 99.0 (NA) — NA indicates that SD could not be calculated for a single participant | 98.6 (1.52)

18. Primary Outcome: Part 2: Absolute Values of Respiration Rate
Description: Respiration rate was measured in semi-supine position after 5 minutes rest
Time Frame: Pre dose, 5 minutes, 15 minutes, 30 minutes, 1 hour and 4 hours post-dose
Population: Safety Population. Only those participants with data available at specified data points were analyzed (represented by n=X in category titles). Participants analysed (25) is greater than the number participants (14) started in Part 2 because Part 2 is a crossover design and participants were considered for 2 dosing sessions.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Breaths per minute
  Pre dose, n=7,5,2,5,1,5 | 16.0 (1.63) | 15.8 (1.64) | 18.0 (1.41) | 14.8 (1.79) | 18.0 (NA) — NA indicates that SD could not be calculated for a single participant | 15.0 (2.00)
  5 minutes, n=7,4,2,5,1,5: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 5
  5 minutes, n=7,4,2,5,1,5 | 15.4 (2.51) | 17.0 (2.16) | 17.0 (2.83) | 15.2 (1.30) | 14.0 (NA) — NA indicates that SD could not be calculated for a single participant | 16.8 (2.28)
  15 minutes, n=7,5,2,5,1,5 | 16.1 (1.86) | 15.6 (1.14) | 15.5 (0.71) | 15.4 (0.55) | 14.0 (NA) — NA indicates that SD could not be calculated for a single participant | 16.6 (2.70)
  30 minutes, n=7,5,2,5,1,5 | 15.6 (1.99) | 15.6 (1.82) | 14.5 (0.71) | 15.0 (1.87) | 14.0 (NA) — NA indicates that SD could not be calculated for a single participant | 15.6 (1.14)
  1 hour, n=7,5,2,5,1,5 | 15.4 (0.79) | 15.6 (1.14) | 15.0 (1.41) | 13.8 (2.05) | 14.0 (NA) — NA indicates that SD could not be calculated for a single participant | 15.6 (0.89)
  4 hours, n=7,5,2,5,1,5 | 16.0 (1.63) | 15.4 (1.34) | 17.5 (0.71) | 15.0 (2.00) | 15.0 (NA) — NA indicates that SD could not be calculated for a single participant | 15.6 (1.52)

19. Primary Outcome: Part 2: Plasma Concentration Time Profile of Oxytocin.
Description: as for outcome 1
Time Frame: -1 hour,-30 minutes,-15 minutes pre-dose, 2 minutes, 3 minutes, 5 minutes, 8 minutes,10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours and 4 hours post dose
Population: Pharmacokinetic Population. Only those participants with data available at specified data points were analyzed (represented by n=X in category titles). Participants analysed (25) is greater than the number participants (14) started in Part 2 because Part 2 is a crossover design and participants were considered for 2 dosing sessions.
Measure: Median (Full Range); unit: Picograms per milliliter
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Picograms per milliliter
  -1 hour; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  -1 hour; n=7, 4, 2, 5, 1, 4 | 0.000 [0.000 to 0.000] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  -30 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  -30 minutes; n=7, 4, 2, 5, 1, 4 | 0.000 [0.000 to 0.000] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  -15 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  -15 minutes; n=7, 4, 2, 5, 1, 4 | 0.000 [0.000 to 0.000] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  2 minutes; n=7, 3, 2, 5, 1, 4: number analyzed (Participants) | 7 | 3 | 2 | 5 | 1 | 4
  2 minutes; n=7, 3, 2, 5, 1, 4 | 114.840 [31.71 to 418.11] | 1081.270 [954.86 to 1166.49] | 219.930 [36.96 to 402.90] | 274.840 [47.89 to 526.82] | 727.660 [727.66 to 727.66] | 284.160 [157.26 to 446.00]
  3 minutes; n=7, 3, 2, 5, 1, 4: number analyzed (Participants) | 7 | 3 | 2 | 5 | 1 | 4
  3 minutes; n=7, 3, 2, 5, 1, 4 | 157.710 [50.71 to 664.51] | 1096.990 [910.90 to 1294.71] | 496.705 [349.05 to 644.36] | 345.610 [83.23 to 655.70] | 1312.740 [1312.74 to 1312.74] | 539.615 [440.78 to 1060.64]
  5 minutes; n=7, 3, 2, 5, 1, 4: number analyzed (Participants) | 7 | 3 | 2 | 5 | 1 | 4
  5 minutes; n=7, 3, 2, 5, 1, 4 | 167.250 [57.34 to 551.96] | 627.240 [504.07 to 812.48] | 697.740 [697.69 to 697.79] | 364.740 [124.40 to 567.33] | 827.940 [827.94 to 827.94] | 622.175 [511.83 to 1309.51]
  8 minutes; n=7, 2, 2, 5, 1, 4: number analyzed (Participants) | 7 | 2 | 2 | 5 | 1 | 4
  8 minutes; n=7, 2, 2, 5, 1, 4 | 145.500 [54.92 to 471.11] | 456.100 [415.88 to 496.32] | 554.120 [515.82 to 592.42] | 287.980 [173.56 to 507.98] | 507.620 [507.62 to 507.62] | 560.665 [522.35 to 899.48]
  10 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  10 minutes; n=7, 4, 2, 5, 1, 4 | 142.900 [62.69 to 407.67] | 345.845 [205.24 to 410.44] | 422.745 [395.49 to 450.00] | 319.960 [189.58 to 416.07] | 431.980 [431.98 to 431.98] | 464.925 [417.84 to 584.43]
  15 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  15 minutes; n=7, 4, 2, 5, 1, 4 | 131.970 [71.72 to 343.15] | 197.855 [157.07 to 206.02] | 228.795 [176.11 to 281.48] | 250.260 [173.25 to 366.23] | 266.140 [266.14 to 266.14] | 234.745 [213.78 to 290.64]
  20 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  20 minutes; n=7, 4, 2, 5, 1, 4 | 128.510 [62.30 to 278.18] | 128.060 [94.91 to 139.29] | 146.675 [108.99 to 184.36] | 230.840 [163.70 to 290.43] | 159.500 [159.50 to 159.50] | 138.780 [130.76 to 176.35]
  30 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  30 minutes; n=7, 4, 2, 5, 1, 4 | 100.500 [57.46 to 183.49] | 63.485 [50.30 to 74.87] | 75.630 [53.02 to 98.24] | 200.950 [130.12 to 211.65] | 80.120 [80.12 to 80.12] | 65.560 [60.35 to 82.21]
  45 minutes; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  45 minutes; n=7, 4, 2, 5, 1, 4 | 54.400 [35.50 to 102.79] | 29.290 [21.05 to 32.88] | 34.125 [22.53 to 45.72] | 133.290 [91.63 to 163.78] | 39.220 [39.22 to 39.22] | 30.945 [21.41 to 33.89]
  1 Hour; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  1 Hour; n=7, 4, 2, 5, 1, 4 | 32.980 [22.90 to 65.79] | 15.095 [11.32 to 21.81] | 22.145 [12.03 to 32.26] | 84.240 [65.27 to 112.31] | 21.290 [21.29 to 21.29] | 15.495 [14.69 to 19.35]
  1.5 Hours; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  1.5 Hours; n=7, 4, 2, 5, 1, 4 | 16.180 [9.74 to 28.43] | 5.580 [4.09 to 1100.01] | 8.170 [4.74 to 11.60] | 41.270 [30.05 to 59.89] | 7.200 [7.20 to 7.20] | 5.160 [4.51 to 6.11]
  2 Hours; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  2 Hours; n=7, 4, 2, 5, 1, 4 | 7.250 [3.66 to 15.40] | 2.885 [2.00 to 19.51] | 2.960 [0.00 to 5.92] | 19.770 [10.73 to 23.97] | 3.500 [3.50 to 3.50] | 2.460 [0.00 to 2.72]
  2.5 Hours; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  2.5 Hours; n=7, 4, 2, 5, 1, 4 | 4.090 [0.00 to 8.86] | 0.000 [0.00 to 73.60] | 0.000 [0.00 to 0.00] | 9.640 [5.41 to 12.03] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  3 Hours; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  3 Hours; n=7, 4, 2, 5, 1, 4 | 2.470 [0.00 to 5.33] | 0.000 [0.00 to 4.11] | 0.000 [0.00 to 0.00] | 5.740 [2.64 to 7.31] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  4 Hours; n=7, 4, 2, 5, 1, 4: number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
  4 Hours; n=7, 4, 2, 5, 1, 4 | 0.000 [0.00 to 2.91] | 0.000 [0.00 to 13.36] | 0.000 [0.00 to 0.00] | 2.910 [0.00 to 4.43] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

20. Primary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Oxytocin
Description: as for outcome 2
Time Frame: as for outcome 19
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed. Participants analysed (23) is greater than the number participants (14) started in Part 2 because Part 2 is a crossover design and participants were considered for 2 dosing sessions.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
Picogram per milliliter | 224.25 (92.5) | 838.25 (67.2) | 697.74 (0.0) | 357.38 (51.4) | 1312.74 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 721.68 (42.2)

21. Primary Outcome: Part 2: Observed Plasma Concentration (Cp)10 of Oxytocin
Description: as for outcome 3
Time Frame: 10 minutes post dose
Population: Pharmacokinetic Population. Participants analysed (25) is greater than the number participants (14) started in Part 2 because Part 2 is a crossover design and participants were considered for 2 dosing sessions.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Picogram per milliliter | 179.98 (79.6) | 293.00 (32.1) | 421.87 (9.1) | 292.95 (37.7) | 431.98 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 407.99 (39.6)

22. Primary Outcome: Part 2: Observed Plasma Concentration (Cp)20 of Oxytocin
Description: as for outcome 3
Time Frame: 20 minutes post dose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Picogram per milliliter | 131.72 (61.1) | 110.44 (26.0) | 141.75 (38.5) | 231.76 (22.2) | 159.50 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 131.21 (25.8)

23. Primary Outcome: Part 2: Observed Plasma Concentration (Cp)30 of Oxytocin
Description: as for outcome 3
Time Frame: 30 minutes post dose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 5 | 2 | 5 | 1 | 5
Picogram per milliliter | 93.54 (49.6) | 56.70 (26.3) | 72.17 (45.8) | 184.71 (20.6) | 80.12 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 63.02 (20.6)

24. Primary Outcome: Part 2: Time to Reach Maximum Observed Concentration (Tmax) of Oxytocin
Description: as for outcome 6
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Median (Full Range); unit: Hours
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
Hours | 0.08333 [0.0500 to 0.2500] | 0.04167 [0.0333 to 0.1833] | 0.0833 [0.0833 to 0.0833] | 0.0833 [0.0500 to 0.3333] | 0.05000 [0.0500 to 0.0500] | 0.08333 [0.0833 to 0.1333]

25. Primary Outcome: Part 2: Area Under the Concentration-time Curve From Time Zero Extrapolated to Time 't' (AUC[0-t]) of Oxytocin
Description: as for outcome 7
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*picogram per milliliter
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 4 | 2 | 5 | 1 | 4
Hour*picogram per milliliter | 127.58 (58.6) | 161.39 (44.1) | 164.46 (15.8) | 247.42 (22.3) | 208.37 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 171.21 (23.9)

26. Primary Outcome: Part 2: Plasma Clearance (CL) of Oxytocin for IV Route Only
Description: Blood samples were collected at indicated time points to evaluate plasma clearance of oxytocin IV bolus and infusion. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 19
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed. Only IV reporting arms presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 3 | 2 | 1 | 4
Liters per hour | 57.93 (46.3) | 50.85 (16.1) | 40.44 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 49.23 (23.6)

27. Primary Outcome: Part 2: Volume of Distribution (VOD) of Oxytocin for IV Route Only
Description: Blood samples were collected at indicated time points to evaluate volume of distribution of oxytocin IV bolus and infusion. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 19
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 3 | 2 | 1 | 4
Liters | 31.22 (56.5) | 25.50 (7.8) | 20.85 (NA) — NA indicates that Geometric Coefficient of Variation could not be calculated for a single participant | 23.47 (27.4)

28. Primary Outcome: Part 2: Time to Reach Terminal Phase Half-life (t1/2) of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate t1/2 of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 19
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed. Participants analysed (22) is greater than the number participants (14) started in Part 2 because Part 2 is a crossover design and participants were considered for 2 dosing sessions.
Measure: Median (Full Range); unit: Hours
Arm/Group | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
Number analyzed (Participants) | 7 | 3 | 2 | 5 | 1 | 4
Hours | 0.5523 [0.376 to 0.882] | 0.3728 [0.341 to 0.411] | 0.3525 [0.294 to 0.411] | 0.6154 [0.422 to 0.721] | 0.357 [0.357 to 0.357] | 0.3398 [0.260 to 0.398]

29. Secondary Outcome: Part 1: Number of Participants With Non-SAEs and SAEs
Description: An adverse event is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function.
Time Frame: Up to 15 days
Population: Safety Population includes participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Participants
  Any non-SAE | 3 | 2
  Any SAE | 2 | 2

30. Secondary Outcome: Part 1: Absolute Values for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: 30 minutes and 2 hours post dose
Population: Safety Population. Only those participants with data available at specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Millimeters of mercury
  SBP: 30 minutes; n=9, 8 | 114.2 (10.35) | 121.5 (19.65)
  SBP: 2 hours; n=9, 7: number analyzed (Participants) | 9 | 7
  SBP: 2 hours; n=9, 7 | 111.0 (16.63) | 110.0 (10.21)
  DBP: 30 minutes; n=9, 8 | 66.2 (5.31) | 69.9 (11.37)
  DBP: 2 hours; n=9, 7: number analyzed (Participants) | 9 | 7
  DBP: 2 hours; n=9, 7 | 65.1 (8.48) | 64.0 (9.04)

31. Secondary Outcome: Part 1: Absolute Values of Heart Rate
Description: Heart rate was measured in semi-supine position after 5 minutes rest
Time Frame: 30 minutes and 2 hours post dose
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Beats per minute
  30 minutes; n= 9, 8 | 86.9 (19.85) | 86.4 (23.05)
  2 hours; n= 9, 7: number analyzed (Participants) | 9 | 7
  2 hours; n= 9, 7 | 86.0 (16.89) | 83.0 (11.27)

32. Secondary Outcome: Part 1: Absolute Values of Respiration Rate
Description: Respiration rate was measured in semi-supine position after 5 minutes rest
Time Frame: 30 minutes and 2 hours post dose
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 7
Breaths per minute
  30 minutes | 14.4 (2.55) | 14.6 (3.15)
  2 hours | 14.7 (2.06) | 14.1 (2.19)

33. Secondary Outcome: Part 1: Absolute Values of Temperature
Description: Body temperature was measured in semi-supine position after 5 minutes rest
Time Frame: 30 minutes and 2 hours post dose
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 7
Degrees Celsius
  30 minutes | 37.29 (0.699) | 36.69 (0.135)
  2 hours | 37.03 (0.581) | 36.90 (0.173)

34. Secondary Outcome: Part 1: Change From Baseline in SBP and DBP
Description: as for outcome 11
Time Frame: Baseline (Day 1, pre-dose), 30 minutes and 2 hours post dose
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Millimeters of mercury
  SBP: 30 minutes; n= 9, 8 | 0.1 (8.39) | 11.4 (17.48)
  SBP: 2 hours; n=9, 7: number analyzed (Participants) | 9 | 7
  SBP: 2 hours; n=9, 7 | -3.1 (13.27) | -0.9 (13.21)
  DBP: 30 minutes; n= 9, 8 | -4.0 (11.14) | -0.1 (13.17)
  DBP: 2 hours; n=9, 7: number analyzed (Participants) | 9 | 7
  DBP: 2 hours; n=9, 7 | -5.1 (10.43) | -6.0 (11.47)

35. Secondary Outcome: Part 1: Change From Baseline in Heart Rate
Description: as for outcome 12
Time Frame: Baseline (Day 1, pre-dose), 30 minutes and 2 hours post dose
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Beats per minute
  30 minutes; n= 9, 8 | 0.2 (16.41) | 4.8 (22.75)
  2 hours; n=9, 7: number analyzed (Participants) | 9 | 7
  2 hours; n=9, 7 | -0.7 (10.39) | 1.9 (9.81)

36. Secondary Outcome: Part 1: Change From Baseline in Respiration Rate
Description: Respiration rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Baseline was defined as the latest pre-dose assessment with a non-missing value at Day 1 (Pre-dose). Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), 30 minutes and 2 hours post dose
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 7
Breaths per minute
  30 minutes | 0.3 (2.12) | -0.3 (2.75)
  2 hours | 0.6 (2.24) | -0.7 (1.89)

37. Secondary Outcome: Part 1: Change From Baseline in Body Temperature
Description: Body temperature was measured at indicated time points in semi-supine position after 5 minutes rest. Baseline was defined as the latest pre-dose assessment with a non-missing value at Day 1 (Pre-dose). Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), 30 minutes and 2 hours post dose
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 7
Degrees Celsius
  30 minutes | 0.60 (0.740) | -0.01 (0.434)
  2 hours | 0.34 (0.623) | 0.20 (0.277)

38. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Three Hours (AUC ([0-3]) of Oxytocin
Description: Blood samples were collected at indicated time points to evaluate AUC (0-3) of oxytocin. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Predose, 3 minutes, 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 2.5 hours and 3 hours post dose on Day 1
Population: Pharmacokinetic Population.
Measure: Mean (Standard Deviation); unit: Hour*picogram per milliliter
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM
Number analyzed (Participants) | 9 | 8
Hour*picogram per milliliter | NA (NA) — NA indicates that data could not be calculated as all values at specified time points (up to 3 hours post-dose) were below the limit of quantification. | NA (NA) — NA indicates that data could not be calculated as all values at specified time points (up to 3 hours post-dose) were below the limit of quantification.

ADVERSE EVENTS:
Time Frame: All non-SAEs and SAEs were collected from start of the study treatment (Day 1) up to Day 15 for Part 1 and up to Day 37 for Part 2.
Description: Non-SAEs and SAEs are reported for Safety Population.
Groups:
- Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus: Healthy participants of childbearing potential receiving oral contraceptive along with 8.5 mcg oxytocin IV bolus. When the duration of IV oxytocin administered was less than or equal to 2 minutes then the IV dose administered was classified as an IV Bolus.
Arm/Group | 400 mcg Oxytocin IH | 17 mcg Oxytocin IM | Combined Oral Contraceptives+400 mcg Oxytocin IH | Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/7 | 0/5 | 0/2 | 0/5 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/8 | 0/7 | 0/5 | 0/2 | 0/5 | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 3/9 | 2/8 | 7/7 | 5/5 | 1/2 | 3/5 | 1/1 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mcg Oxytocin IH (N=9) | 17 mcg Oxytocin IM (N=8) | Combined Oral Contraceptives+400 mcg Oxytocin IH (N=7) | Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus (N=5) | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion (N=2) | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH (N=5) | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus (N=1) | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion (N=5)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mcg Oxytocin IH (N=9) | 17 mcg Oxytocin IM (N=8) | Combined Oral Contraceptives+400 mcg Oxytocin IH (N=7) | Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus (N=5) | Combined Oral Contraceptives+ 8.5 mcg Oxytocin IV Infusion (N=2) | Non-Combined Oral Contraceptives+400 mcg Oxytocin IH (N=5) | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Bolus (N=1) | Non-Combined Oral Contraceptive+ 8.5 mcg Oxytocin IV Infusion (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02999100/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT02999100/SAP_001.pdf